CLINICAL TRIAL: NCT02379715
Title: Effect-site Concentration of Remifentanil for Smooth Induction With Desflurane
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, clinical assistant professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-MED-CT4-14-327
Record Dates: First submitted 2015-01-27; First posted 2015-03-05 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia
Keywords: Remifentanil; smooth induction; desflurane
MeSH Terms: interventions — Remifentanil; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remifentanil (Experimental): When the particapants arrived into the operating room, the investigators applied standard monitoring and after preoxygenation, 2 mg remifentanil was diluted into 50 ml of normal saline (40 μg/ml solution) and was infused by Target concentration infusion (TCI) via syringe pump (Pilot Anesthesia 2. Fresenius vial, France) using the pharmacokinetic model. Investigator started to infuse remifentanil at 4 ng/ml and after the Ce of remifentanil reached the target concentration level, opened the dial of desflurane vaporizer at 4 vol%. After 30 seconds, increase the concentration of desflurane 8% and 12% at last. If there is no spontaneous respiration or loss of consciousness, the muscle relaxant esmerone 0.6mg/kg is injected and after 90 seconds the tracheal intubation is performed.
  Interventions: Drug: Remifentanil; Drug: Desflurane

INTERVENTIONS:
Drug: Remifentanil
  Other Names: Ultiva
Drug: Desflurane

SUMMARY:
Desflurane is a halogenated ether with low solubility, giving rapid induction and emergence from anesthesia This character is suitable for Volatile Induction and Maintenance Anesthesia (VIMA). But desflurane can cause airway irritation when it used as a sole induction agent to adult or children, so there were many studies about reducing the airway reflex combined with desflurane.

Remifentanil is a short acting opioid and is quickly hydrolyzed by nonspecific esterase in the plasma and multiorgan. Several studies suggest the optimal dose of remifentanil for reducing airway reflex or cardiovascular response for intubation combined with desflurane. But these studies were under 1 Minimal Alveolar Concentration (MAC) of desflurane and this point could be a limitation because desflurane concentration over 1 MAC increase airway irritation significantly. This study this study was designed to determine a median effective effect-site concentration (EC50) of remifentanil to prevent airway irritation during desflurane anesthesia over 1 MAC.

ELIGIBILITY:
Inclusion Criteria:

* patients for surgery requiring general anesthesia
* American Society of Anesthesiologists(ASA) classification I, II

Exclusion Criteria:

* history of gastroesophageal reflux, High grade obesity, Predicted difficult airway, Asthma, Chronic obstructive pulmonary disease(COPD), Upper respiratory infection (URI) within 3 weeks

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Fail or success for induction with desflurane | After loss of consciousness, 5 seconds
  Failure for induction with desflurane is defined if there is a cough, laryngospasm, hypoxia or any refusal movement of patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yoonjeong Chae, MD, Study Chair — Ajou University School of Medicine